CLINICAL TRIAL: NCT04089826
Title: Role of LTOT in Pateints With ILD
Brief Title: Long Term Oxygen Therapy in Patients With Interstitial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Mohammed Eltayeb, Resident at chest department Assiut university, Assiut University
Other Study IDs: Role of LTOT in Pateints e ILD
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Long Term Oxygen Therapy; Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the effect of using long term oxygen therapy in patients with interstitial lung disease and chronic hypoxia

DETAILED DESCRIPTION:
long term oxygen can be used in patients with interstitial lung disease with hypoxia and the aim of this study is to k ow whether this will improve life style , exercise tolerance in those patients

ELIGIBILITY:
Inclusion Criteria :

* patients with ILD and hypoxia with SO2<88 at room air and PO2 < or equal 7.3k.pa or < or equal 8 k.pa in presence of lower limb edema , pulmonary hypertension or polycythemia
* age group 18 : 70

Exclusion Criteria :

* Causes of chronic respiratory failure other than ILD.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with ILDs who are prescribed for LTOT between eighteen and seventy years old
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Dyspnea score improvement | Baseline
  dyspnea by Modified Medical Research Counsel
Quality of life improvement | Baseline
  Quality of life by st.George questionnaire

REFERENCES:
- [Background] Cobo-Ibanez T, Lopez-Longo FJ, Joven B, Carreira PE, Munoz-Fernandez S, Maldonado-Romero V, Larena-Grijalba C, Cubas IL, Muriel ET, Mateos CB, de la Pena Lefebvre PG, Gomez-Gomez A, Nogal LB, Perez A, Almodovar R, Lojo L, Ruiz-Gutierrez L, Lopez-Robledillo JC, Garcia de Yebenes MJ, Nuno-Nuno L. Long-term pulmonary outcomes and mortality in idiopathic inflammatory myopathies associated with interstitial lung disease. Clin Rheumatol. 2019 Mar;38(3):803-815. doi: 10.1007/s10067-018-4353-2. Epub 2018 Nov 3. PMID 30392161